CLINICAL TRIAL: NCT07039214
Title: The Relationship of Thoracolumbar Fascia Flexibility With Trunk Proprioception and Spinal Posture in Individuals With Non-specific Low Back Pain
Brief Title: Thoracolumbar Fascia Flexibility and Trunk Proprioception Relationship With Spinal Posture
Status: Completed | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ramazan KURUL, Assist. Prof, Abant Izzet Baysal University
Other Study IDs: AIBU-FTR-RK-10
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Low Back Pain, Mechanical
Keywords: Proprioception; Fascia
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-Specific low back pain group: Patients with non-Specific low back pain was included in this group.
  Interventions: Other: Observation of low-back pain symptoms
- Asymptomatic group: Healthy people with no low back pain or any other symptom related to this region.
  Interventions: Other: Observation of healthy comparators

INTERVENTIONS:
Other: Observation of low-back pain symptoms — No intervention was applied.
  Groups: Non-Specific low back pain group
Other: Observation of healthy comparators — No intervention was applied.
  Groups: Asymptomatic group

SUMMARY:
This study aimed to examine the associations between thoracolumbar fascia flexibility, trunk proprioception, and spinal posture in individuals experiencing non-specific low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to voluntarily participate in the study
* Age range between 35 and 65 years
* Reporting a pain intensity in the lumbar region greater than 3 on the Visual Analog Scale (VAS)
* Experiencing lumbar region pain for a duration of at least three months
* Reporting pain intensity below 3 on the VAS in any other part of the body

Exclusion Criteria:

* History of surgical intervention in the lumbar region
* Being diagnosed with conditions such as osteoporosis, rheumatic diseases infection, fracture, structural deformity, cauda equina syndrome, tumor, radicular syndrome, or inflammatory disorders
* Classification as "very active" based on the International Physical Activity Questionnaire (IPAQ) criteria
* Hypermobility, defined as a Beighton Score of 4 or higher
* Pregnancy

Ages: 35 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with non-specific low back pain and healthy participants of same age were included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Thoracolumbar fascia flexibility | baseline
  The goniometric platform will be placed on a table in front of the participants to measure thoracolumbar flexibility (TLF). Participants will be seated on an unsupported chair with the lumbar region in a neutral position and the knees and hips flexed at 90°. The pelvis will be stabilized by the researcher holding the spina iliaca posterior superior. Participants will be instructed to rotate their trunk first to the right and then to the left, following verbal cues provided by the researcher. At the endpoint of each rotation, participants will be asked to mark the platform in front of them while maintaining 90° shoulder flexion, with their hands clasped in front of the trunk and holding a wooden pen between their hands. Each measurement will be performed three times for each side, and the average value will be recorded.

SECONDARY OUTCOMES:
Proprioception Measurement | baseline
  The "Clinometer" mobile application will be used to assess proprioception. Participants will stand upright with their arms at their sides, heels spaced 3 cm apart, and their gaze fixed on a point at eye level. The phone will be placed in an upright position just above the iliac crest, aligned with the mid-axillary line at the midpoint of the iliac spine, and secured with a belt. The inclination of the clinometer will be calibrated to 0°, which will serve as the starting point. The range of motion will be limited to 0-30°.
  The physiotherapist will first passively move the participant's trunk to the target angle, where the participant will remain for 10 seconds to memorize the position. Afterward, the participant will actively return to the starting position. Then, the participant will be instructed to actively replicate the target angle three times with their eyes closed. The mean deviation across the three attempts will be recorded as the proprioception value.
Spinal Posture Assessment | baseline
  The Spinal Mouse (Idiag, Voletswil, Switzerland, SM) device will be employed to assess spinal posture. Prior to the measurement, the researcher will demonstrate all required positions to the participants. Participants will be instructed to hold each position for 1-2 seconds. They will be asked to remove their clothing to expose all spinous processes, which will be palpated and marked from C7 to S3 using a felt-tip pen by the researcher. The Spinal Mouse will then be guided along the marked points from top to bottom.
  Participants will be evaluated in three positions: upright, maximum trunk flexion, and maximum trunk extension.
Visual Analog Scale | baseline
  Pain intensity will be assessed using a 0-10 cm horizontal Visual Analog Scale (VAS). On this scale, a 10 cm line will be anchored with "0: no pain" at one end and "10: unbearable pain" at the other. Participants will be instructed to indicate the intensity of their pain by placing a dot, drawing a line, or marking a specific point along the scale. The distance from the starting point to the participant's mark will represent their perceived pain intensity. Pain levels will be classified as follows: 0-3.4 cm will indicate mild pain, 3.5-7.4 cm moderate pain, and 7.5 cm or more severe pain.
Oswestry Low Back Pain Disability Questionnaire | baseline
  The Oswestry Disability Questionnaire will be widely utilized to assess specific outcomes in individuals with spinal problems. It will consist of 10 items that evaluate various functional aspects, each scored on a scale from 0 to 5. The total score will be calculated by summing the individual item scores, multiplying the result by 2, and expressing it as a percentage. Higher percentages will indicate greater levels of disability.
  Scoring classifications will be as follows:
  0-20%: Low back pain will not significantly impact the individual's daily life.
  20-40%: Low back pain will mildly restrict the individual's daily activities.
  40-60%: Low back pain will severely restrict the individual's daily activities.
  60-80%: The individual's daily life will be significantly impaired due to low back pain.
  80-100%: The individual will be considered bedridden (symptoms may be exaggerated).
International Physical Activity Questionnaire - Short Form | baseline
  This questionnaire will be a standardized tool developed by researchers from multiple countries, supported by the World Health Organization, to assess levels of physical activity. The original version will consist of 27 items, while the short form will include 7 items. Participants will be asked to estimate the duration and frequency of their physical activity over the previous week. The reported durations will be multiplied by known metabolic equivalents values for each activity, and an overall score will be calculated by summing the results for all items. Scores for walking, moderate activity, and vigorous activity will be determined by summing the corresponding item scores. Time spent sitting will be excluded from the calculation.

CONTACTS AND LOCATIONS:
Overall Officials: ramazan kurul, Ph.D, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Faculty of Health Sciences Bolu Abant Izzet Baysal University, Bolu, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No